CLINICAL TRIAL: NCT06208046
Title: Machine Learning Models to Predict 5-Year Post-Surgery Survival of Older Gastric Cancer Patients
Brief Title: Predict 5-Year Survival in Elderly Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Collaborators: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Other Study IDs: 2023KY237
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer; Machine Learning
Keywords: Gastric Cancer; Elderly; Oxidative Stress; Machine Learning; Overall Survival
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, elderly patients with gastric cancer who underwent radical gastrectomy in Union Hospital Affiliated to Fujian Medical University from 2012 to 2018 were included as a derived cohort, and the training set and internal validation set were randomly divided by 4:1. Machine learning strategies of random forest, decision tree and support vector machine are used to construct survival prediction model. Each model was tested in an internal validation set and an external validation set consisting of patients from two other large medical centers.

DETAILED DESCRIPTION:
This is a retrospective, supervised learning, data mining study.

ELIGIBILITY:
Inclusion Criteria:

* (1) GC diagnosis confirmed by abdominal computed tomography (CT) or biopsy; (2) age ≥65 years at diagnosis; (3) underwent radical surgical resection without evidence of distant metastasis; and (4) availability of complete clinical and pathological data.

Exclusion Criteria:

* (1) postoperative pathology confirming non-gastric primary tumors; (2) distant metastasis; (3) incomplete clinical data; and (4) other concurrent malignancies within five years.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This retrospective prognostic study encompassed patients aged 65 or older who underwent radical gastrectomy for GC from January 2012 to April 2018. The study involved a derivation cohort and an external validation cohort.
Sampling Method: Non-Probability Sample
Enrollment: 2187 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
5-year overall survival | 5 years or 60 months.
  Survival status at 5 years: survival, death, survival with tumor, deletion.

CONTACTS AND LOCATIONS:
Overall Officials: Huang Chang-Ming, Prof., Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Zhang XQ, Huang ZN, Wu J, Zheng CY, Liu XD, Huang YQ, Chen QY, Li P, Xie JW, Zheng CH, Lin JX, Zhou YB, Huang CM. Development and validation of a prognostic prediction model for elderly gastric cancer patients based on oxidative stress biochemical markers. BMC Cancer. 2025 Feb 1;25(1):188. doi: 10.1186/s12885-025-13545-x. PMID 39893402